CLINICAL TRIAL: NCT02934997
Title: The Role of Dysfunctional HDL in Community and Hospital Acquired Sepsis
Brief Title: The Role of Dysfunctional HDL in Sepsis
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201701349-N; UFlorida (Other: University of Florida); 1K23GM115690-01 (NIH); UFJ2016-032 (Other: University of Florida, Jacksonville)
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Sepsis; Septic Shock
Keywords: sepsis; septic shock; cholesterol; high density lipoprotein
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of Serum and Plasma will be drawn and retained for several clinically relevant biomarkers as well as future testing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Community-Acquired Sepsis: The Adult ED at UF JAX is a high volume, high acuity ED which treats approximately 90,000 patients per year. All CA-sepsis patients will be recruited from the UF JAX ED. Patients meeting the recently updated definition of sepsis (suspected or confirmed infection plus ≥ 2 SOFA points) OR septic shock (hypotension not responsive to 30 mL/kg IV fluids, vasopressor requirement, and lactate ≥ 2) and being treated with an institutional, evidence-based guideline (EBG) management bundle for sepsis within 24 hours presenting to the UF Health Jacksonville Emergency Department (ED) will be approached for enrollment.
  Interventions: Other: Observational study
- Hospital-Acquired Sepsis: UFH (Gainesville) is a Level 1 Trauma Center and surgical tertiary care center with 24 trauma intensive care unit (ICU) and 24 surgery ICU beds and are the primary ICUs for almost every surgical patient in the hospital and the location for recruitment for Project #1 of the Sepsis P50. Patients meeting the recently updated definition of sepsis (suspected or confirmed infection plus ≥ 2 SOFA points) OR septic shock (hypotension not responsive to 30 mL/kg IV fluids, vasopressor requirement, and lactate ≥ 2) and being treated with an institutional, evidence-based guideline (EBG) management bundle for sepsis within 24 hours in the UFH Surgical ICU will be approached for enrollment.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study

SUMMARY:
To determine the role of dysfunctional high density lipoprotein (Dys-HDL) in predicting or mediating progression to chronic critical illness or morbid long-term outcomes in patients being treated for community-acquired or hospital-acquired sepsis.

DETAILED DESCRIPTION:
The long-term goal of this research program is to characterize the antecedents and mediators of morbid long-term outcomes in patients with sepsis. Despite successful early management, sepsis is a disease with a high incidence of chronic critical illness (CCI - intensive care unit stay ≥ 14 days with organ dysfunction) and morbid long-term outcomes (functional dependence or death at 1 year), which occur frequently in early survivors. Both the rapid identification of patients at risk for morbid outcomes and the development of novel therapies are crucial for improving outcomes after sepsis. High density lipoprotein (HDL) defends against sepsis-associated organ injury by: 1) neutralizing bacterial endotoxin, 2) modulating innate cellular immunity and preventing release of inflammatory cytokines, and 3) preventing endothelial cell activation and dysfunction. However, HDL can become dysfunctional (Dys-HDL) in the setting of inflammation, losing protective functions and becoming pro-inflammatory. Our preliminary results demonstrate that Dys-HDL is present in early sepsis and that persistent Dys-HDL elevation (first 48 hours) is associated with adverse outcomes (death, hospice or nursing home care). The overall goal of this proposal is to investigate and fully characterize the role of Dys-HDL in a diverse population of patients with both CA and HA-sepsis. The central hypothesis of this study is that structural and functional changes in HDL during sepsis are associated with the persistent presence of Dys-HDL as well as the inflammation and endothelial dysfunction that lead to acute organ dysfunction, CCI, and morbid long-term outcomes. To test this, we will enroll 160 patients in a two-site, prospective, longitudinal, cohort study.

ELIGIBILITY:
Inclusion Criteria:

* patients meeting the recently updated definition of sepsis (suspected or confirmed infection plus ≥ 2 SOFA points) OR septic shock (hypotension not responsive to 30 mL/kg IV fluids, vasopressor requirement, and lactate ≥ 2)23 and being treated with an institutional, evidence-based guideline (EBG) management bundle for sepsis within 24 hours which has been adopted at both sites.

Exclusion Criteria:

* significant traumatic brain injury (evidence of neurologic injury on CT scan and a GCS <8)
* refractory shock (likely death within 12 hours)
* alternative/confounding diagnosis causing shock (e.g., myocardial infarction or pulmonary embolus)
* uncontrollable source of sepsis (e.g., irreversible disease state such as unresectable dead bowel)
* patients deemed futile care or have advanced directives limiting resuscitative efforts
* severe CHF (NY Heart Association Class IV)
* Child-Pugh Class B or C liver disease
* HIV/AIDS causing severe immunocompromise
* organ transplant recipient on immunosuppressive agents
* known pregnancy
* inability to obtain informed consent
* diagnosed disorders of lipid metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis or septic shock presenting to both sites.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Early sepsis-associated organ dysfunction, incidence of chronic critical illness and morbid long-term outcomes after sepsis. | 1 year

SECONDARY OUTCOMES:
The temporal relationship between Dys-HDL and sepsis and endothelial biomarkers in patients with sepsis. | 4 days
Explore changes in HDL function from patients with sepsis with rapid recovery versus patients with sepsis who develop CCI versus healthy controls. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Faheem Guirgis, MD, Principal Investigator — University of Florida

REFERENCES:
- [Derived] Labilloy G, Tanaka S, Black LP, Augustin B, Hopson C, Bethencourt J, Wu D, Sulaiman D, Bertrand A, Salomao R, Graim K, Datta S, Reddy S, Guirgis FW, Hofmaenner DA. IDENTIFYING A SEPSIS SUBPHENOTYPE CHARACTERIZED BY DYSREGULATED LIPOPROTEIN METABOLISM USING A SIMPLIFIED CLINICAL DATA ALGORITHM. Shock. 2025 Aug 1;64(2):218-225. doi: 10.1097/SHK.0000000000002605. Epub 2025 Apr 23. PMID 40267485
- [Derived] Augustin B, Wu D, Black LP, Bertrand A, Sulaiman D, Hopson C, Jacob V, Shavit JA, Hofmaenner DA, Labilloy G, Smith L, Cagmat E, Graim K, Datta S, Reddy ST, Guirgis FW. Multiomic molecular patterns of lipid dysregulation in a subphenotype of sepsis with higher shock incidence and mortality. Crit Care. 2024 Dec 24;28(1):431. doi: 10.1186/s13054-024-05216-3. PMID 39716214
- [Derived] Black LP, Hopson C, Barker G, Munson T, Henson M, Bertrand A, Daly-Crews K, Reddy ST, Guirgis FW. TRENDS IN CHOLESTEROL AND LIPOPROTEINS ARE ASSOCIATED WITH ACUTE RESPIRATORY DISTRESS SYNDROME INCIDENCE AND DEATH AMONG SEPSIS PATIENTS. Shock. 2024 Feb 1;61(2):260-265. doi: 10.1097/SHK.0000000000002295. Epub 2023 Dec 28. PMID 38407817